CLINICAL TRIAL: NCT00006018
Title: Phase I Study of BMS-214662 and Paclitaxel in Patients With Advanced Malignancies
Brief Title: Paclitaxel and BMS-214662 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU4Y99; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-4Y99; NCI-290
Record Dates: First submitted 2000-07-05; First posted 2004-03-08 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 7-cyano-2,3,4,5-tetrahydro-1-(1H-imidazol-4-ylmethyl)-3-(phenylmethyl)-4-(2-thienylsulfonyl)-1H-1,4-benzodiazepine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BMS-214662 — This is a dose-escalation study of BMS-214662. BMS-214662 IV over 1 hour on day 3 of course 1. For all subsequent courses, patients receive BMS-214662 IV over 1 hour on day 1 (30 minutes after paclitaxel). Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.
Drug: paclitaxel — Patients receive paclitaxel IV over 3 hours on day 1 of course 1. For all subsequent courses, patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of paclitaxel and BMS-214662 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of BMS-214662 in combination with paclitaxel in patients with advanced solid tumors. II. Determine the safety and tolerability of this regimen in these patients. III. Determine the pharmacokinetics of this treatment regimen in this patient population. IV. Determine the pharmacodynamic effects of this treatment regimen in serial tumor biopsies in these patients. V. Determine the cytotoxicity of this treatment regimen in these patients.

OUTLINE: This is a dose-escalation study of BMS-214662. Patients receive paclitaxel IV over 3 hours on day 1 and BMS-214662 IV over 1 hour on day 3 of course 1. For all subsequent courses, patients receive paclitaxel IV over 3 hours followed 30 minutes later by BMS-214662 IV over 1 hour on day 1. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or objectively responding disease receive additional therapy at the investigator's discretion. Cohorts of 3-6 patients receive escalating doses of BMS-214662 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Patients are followed every 4 weeks.

PROJECTED ACCRUAL: A maximum of 18-21 patients will be accrued for this study within 12-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed solid tumor unresponsive to standard therapy or for which no effective therapy exists Measurable or evaluable disease amenable to CT-guided or percutaneous needle biopsy No active symptomatic brain metastases requiring steroids, including evidence of cerebral edema on CT scan or MRI or progression from prior imaging study

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL ALT/AST no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No history of clinically significant cardiac arrhythmia that could be exacerbated by QT interval prolongation No uncontrolled or significant cardiovascular disease No myocardial infarction within the past 6 months No significant congestive heart failure No second- or third- degree heart block No prolonged QTc interval (greater than 450 ms) on EKG Pulmonary: No uncontrolled or significant pulmonary disease Other: No serious uncontrollable medical disorder or active infection that would preclude study No dementia or altered mental status that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: No more than 2 prior chemotherapy regimens Prior taxanes allowed At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics No concurrent antineoplastic hormonal therapy Concurrent hormone replacement therapy allowed Radiotherapy: At least 4 weeks since prior wide-field radiotherapy No concurrent radiotherapy Surgery: Not specified Other: At least 4 weeks since prior investigational drugs At least 7 days since prior substrates of cytochrome P450-3A4 (CYP3A4) No other concurrent experimental anticancer medications No concurrent dolasetron or droperidol No medications or other agents known to prolong the QT interval for at least 4 half-lives prior to, during, and for 24 hours after administration of BMS-214662 Concurrent antihistamines allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2000-07; Primary Completion 2001-12 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of BMS-214662 in combination with paclitaxel. | Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ireland Cancer Center at University Hospitals Case Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio